CLINICAL TRIAL: NCT03287908
Title: A Phase 1/2 Open-label Study Evaluating the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics, and Efficacy of AMG 701 Monotherapy, or in Combination With Pomalidomide, With and Without Dexamethasone in Subjects With Relapsed or Refractory Multiple Myeloma (ParadigMM-1B)
Brief Title: A Study to Assess AMG 701 Montherapy, or in Combination With Pomalidomide, With or Without, Dexamethasone in Subjects With Relapsed or Refractory Multiple Myeloma
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: business decision, not safety reasons.
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 20170122; 2017-001997-41 (EudraCT Number)
Record Dates: First submitted 2017-09-06; First posted 2017-09-19 (Actual); Last update posted 2025-10-08 (Actual); Status verified 2025-10

CONDITIONS: Relapsed/Refractory Multiple Myeloma
Keywords: Amgen; Phase 1; Phase 2; Phase 1/2; Clinical Trial; Oncology/Hematology; Relapsed/Refractory Multiple Myeloma; Immunotherapy
MeSH Terms: conditions — Multiple Myeloma; Neoplasms | interventions — pomalidomide; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- AMG 701 (Experimental)
  Interventions: Drug: AMG 701
- AMG 701 + Pomalidomide (Experimental)
  Interventions: Drug: AMG 701; Drug: Pomalidomide
- AMG 701 + Pomalidomide + Dexamethasone (Experimental)
  Interventions: Drug: AMG 701; Drug: Pomalidomide; Drug: Dexamethasone

INTERVENTIONS:
Drug: AMG 701 — Subjects will receive IV infusions of AMG 701.
Drug: Pomalidomide — Subjects will receive oral capsules of pomalidomide.
  Arms: AMG 701 + Pomalidomide; AMG 701 + Pomalidomide + Dexamethasone
Drug: Dexamethasone — Subjects will receive IV injections or oral dexamethasone.
  Arms: AMG 701 + Pomalidomide + Dexamethasone

SUMMARY:
The primary purpose of the phase 1 part of the study is to evaluate safety and tolerability of AMG 701 monotherapy to identify the RP2D for AMG 701 monotherapy followed by a dose-confirmation part to gather further safety data for AMG 701 monotherapy at the RP2D in adult subjects with relapsed/refractory multiple myeloma (RRMM). In addition, this study will include a sequential dose exploration part to identify the RP2D of AMG 701 in combination with pomalidomide, with and without dexamethasone (AMG 701-P+/-d). Phase 2 will consist of the dose-expansion part to gain further efficacy and safety experience with AMG 701 monotherapy in adult subjects with RRMM.

ELIGIBILITY:
Inclusion Criteria:

* Multiple myeloma meeting the following criteria:

  * Pathologically-documented diagnosis of multiple myeloma that is relapsed or is refractory as defined by the following:

    * Relapsed after > or = 3 lines of prior therapy that must include all approved and available therapies deemed eligible by the investigator, inclusing at a minimum of a proteasome inhibitor (PI), an immunomodulatory drug (IMiD), and, where approved and available, a CD38-directed cytolytic antibody in combination in the same line or separate lines of treatment OR refractory to PI, IMiD, and CD38- directed cytolytic antibody,
    * Subjects who could not tolerate a PI, IMiDs, or a CD38-directed cytolytic antibody are eligible to enroll in the study.
  * Measurable disease as per IMWG response criteria
* Eastern Cooperative Oncology Group (ECOG) Performance Status of ≤ 2

Inclusion criteria specific to AMG 701-P±d include:

* Subjects must have received ≥ 2 lines of prior therapy that must include a proteasome inhibitor (PI), lenalidomide, and where approved and available a CD38-directed antibody. These therapies may be in the same line or separate lines of treatment.
* Subjects must have responded to at least 1 prior line with at least a PR.
* Subjects that have previously received pomalidomide must not have been removed from therapy due to toxicity attributable to pomalidomide and must be at least 6 months from their last dose of pomalidomide.
* Subjects must not have known intolerance to doses of dexamethasone up to 40 mg weekly (20 mg weekly if > 75 years).

Exclusion Criteria:

* Known extramedullary relapse in the absence of any measurable medullary involvement
* Known central nervous system involvement by multiple myeloma
* Autologous stem cell transplantation less than 90 days prior to study day 1
* Recent history of primary plasma cell leukemia (within last 6 months prior to enrollment) or evidence of primary or secondary plasma cell leukemia at the time of screening
* Waldenstrom's macroglobulinemia
* Prior amyloidosis (subjects with multiple myeloma with asymptomatic deposition of amyloid plaques found on biopsy would be eligible if all other criteria are met)
* Treatment with systemic immune modulators including, but not limited to, nontopical systemic corticosteroids (unless the dose is ≤ 10 mg/day prednisone or equivalent), cyclosporine, and tacrolimus within 2 weeks before study day 1
* Last anticancer treatment (chemotherapy, IMiD, PI, molecular targeted therapy) < 2 weeks prior to study day 1 or treatment with a therapeutic antibody less than 4 weeks prior to study day 1 as well as systemic radiation therapy within 28 days prior to study day 1 or focal radiotherapy within 14 days prior to study day 1.
* Prior treatment with any drug or construct that targets BCMA on tumor cells (eg, other bispecific antibody constructs, antibody drug conjugates, or CAR-T cells), other than Group C where prior treatment with GSK2857916 (belantamab mafodotin) is required.

Exclusion criteria specific to AMG 701-P±d include:

* History of serious hypersensitivity associated with thalidomide, pomalidomide, or lenalidomide (> grade 3).
* Multiple myeloma with IgM subtype.
* POEMS syndrome (polyneuropathy, organomegaly, endocrinopathy, monoclonal protein, and skin changes).
* Contraindication to pomalidomide or dexamethasone.
* Glucocorticoid therapy within 14 days prior to randomization that exceeds a cumulative dose of 160 mg of dexamethasone or equivalent dose of other corticosteroids.
* Treatment with systemic immune modulators including, but not limited to, non-topical systemic corticosteroids (unless the dose is ≤ 10 mg/day prednisone or equivalent), cyclosporine, and tacrolimus within 2 weeks before study day 1 or 4 weeks before study day 1 for Phase 1 dose-confirmation.
* Female subjects of childbearing potential with a positive pregnancy test assessed within 14 days prior to first dose of study drugs and/or a positive urine pregnancy test within 24 hours prior to first dose. In addition, females of childbearing potential unwilling to undergo pregnancy testing weekly during the first 4 weeks of pomalidomide use followed by pregnancy testing every 4 weeks in females with regular menses or every 2 weeks in females with irregular menstrual cycles.
* Male subjects with a female partner of childbearing potential and female subjects of childbearing potential who are unwilling to use 2 methods of contraception (1 of which must be highly effective during the study and for an additional 75 days (females) and 135 days (males) after receiving the last dose of AMG 701, or 28 days after the last dose pomalidomide (males and females) or dexamethasone (females), whichever occurs later.
* Females who are lactating/breastfeeding or who plan to breastfeed while on study through 75 days after receiving the last dose of AMG 701, or 28 days after the last dose pomalidomide or dexamethasone, whichever occurs later.
* Females planning to become pregnant while on study through 75 days after receiving the last dose of AMG 701 or 28 days after the last dose pomalidomide or dexamethasone, whichever occurs later.
* Male subjects with a pregnant partner who are unwilling to practice abstinence or use a latex or synthetic condom (even if they have had a vasectomy with medical confirmation of surgical success) during treatment (including during dose interruptions) and for an additional 135 days after the last dose of AMG 701, or 28 days after the last dose pomalidomide, whichever occurs later.
* Males who are unwilling to abstain from sperm donation while on study through 135 days after receiving the last dose of AMG 701 or 28 days after the last dose pomalidomide, whichever occurs later.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 174 (Actual)
Dates: Start 2017-11-13 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Number of subjects with dose-limiting toxicities (DLTs) | 28 days
Number of subjects with treatment emergent adverse events (TEAEs) | 60 months
Number of subjects with treatment-related adverse events | 60 months
Number of subjects with disease-related adverse events | 60 months
Number of subjects with clinically-significant changes in vital signs | 48 months
Number of subjects with clinically-significant changes in physical examination measurements | 48 months
Number of subjects with clinically-significant changes in electrocardiogram (ECG) measurements | 48 months
Number of subjects with clinically-significant changes in clinical laboratory tests | 48 months

SECONDARY OUTCOMES:
Pharmacokinetic parameter of AMG 701: Maximum concentration (Cmax) | 12 weeks
Pharmacokinetic parameter of AMG 701: Time of maximum concentration (Tmax) | 12 weeks
Pharmacokinetic parameter of AMG 701: Area under the concentration-time curve (AUC) | 12 weeks
Pharmacokinetic parameter of AMG 701: Steady state concentration (Css) | 12 weeks
Anti-tumor activity: Overall response rate | 48 months
  Efficacy parameter measured by International Myeloma Working Group (IMWG) response criteria. Best overall response of stringent CR (sCR), complete response (CR), very good partial response (VGPR), or partial response (PR).
Anti-tumor activity: Best overall response of stringent complete response (sCR) | 48 months
  Efficacy parameter measured by International Myeloma Working Group (IMWG) response criteria.
Anti-tumor activity: Best overall response of complete response (CR) | 48 months
  Efficacy parameter measured by International Myeloma Working Group (IMWG) response criteria.
Anti-tumor activity: Best overall response of very good partial response (VGPR) | 48 months
  Efficacy parameter measured by International Myeloma Working Group (IMWG) response criteria.
Anti-tumor activity: Best overall response of partial response (PR) | 48 months
  Efficacy parameter measured by International Myeloma Working Group (IMWG) response criteria.
Anti-tumor activity: Duration of response | 48 months
  Efficacy parameter measured by International Myeloma Working Group (IMWG) response criteria. Defined as time from the first PR or better to disease progression or death.
Anti-tumor activity: Time to response | 48 months
  Efficacy parameter measured by International Myeloma Working Group (IMWG) response criteria.
Anti-tumor activity: Progression-free survival | 48 months
  Efficacy parameter measured by International Myeloma Working Group (IMWG) response criteria. Defined as time from start of treatment until disease progression or death.
Anti-tumor activity: Overall survival | 60 months
  Defined as time from start of treatment until death due to any cause.
Anti-tumor activity: Number of subjects with minimum residual disease negative complete response | 48 months
  Efficacy parameter measured by International Myeloma Working Group (IMWG) response criteria.
Pharmacokinetic parameter of AMG 701: Trough concentration (Ctrough) | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (34):
- United States (17):
  - Mayo Clinic - Arizona, Scottsdale, Arizona
  - University of Arkansas for Medical Sciences Myeloma Institute Slot 816, Little Rock, Arkansas
  - Mayo Clinic Florida, Jacksonville, Florida
  - Winship Cancer Institute Emory U, Atlanta, Georgia
  - University of Chicago Medical Center - Multiple Myeloma Research Consortium, Chicago, Illinois
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - Washington University, St Louis, Missouri
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Icahn School of Medicine at Mount Sinai, Hackensack, New Jersey
  - Columbia University Medical Center, New York, New York
  - New York Presbyterian Hospital, Weill Cornell Medical College, New York, New York
  - Levine Cancer Institute, Charlotte, North Carolina
  - Wake Forest Baptist Health, Winston-Salem, North Carolina
  - University of Texas MD Anderson Cancer Center, Houston, Texas
  - University of Utah Huntsman Cancer Institute, Salt Lake City, Utah
  - The Medical College of Wisconsin, Milwaukee, Wisconsin
- Australia (3):
  - Princess Alexandra Hospital, Woolloongabba, Queensland
  - Peter MacCallum Cancer Centre, Melbourne, Victoria
  - The Alfred Hospital, Melbourne, Victoria
- Canada (2):
  - University Health Network-Princess Margaret Cancer Centre, Toronto, Ontario
  - McGill University Health Centre Glen Site, Montreal, Quebec
- Germany (3):
  - Universitätsklinikum Heidelberg, Heidelberg
  - Universitätsklinikum Schleswig Holstein Campus Kiel, Kiel
  - Universitaetsklinikum Wuerzburg, Würzburg
- Japan (6):
  - Nagoya City University Hospital, Nagoya, Aichi-ken
  - Gunma University Hospital, Maebashi, Gunma
  - Kobe City Medical Center General Hospital, Kobe, Hyōgo
  - Kanazawa University Hospital, Kanazawa, Ishikawa-ken
  - National Hospital Organization Okayama Medical Center, Okayama, Okayama-ken
  - The Cancer Institute Hospital of Japanese Foundation for Cancer Research, Koto-ku, Tokyo
- Netherlands (3):
  - Universitair Medisch Centrum Groningen, Groningen
  - Maastricht Universitair Medisch Centrum, Maastricht
  - Universitair Medisch Centrum Utrecht, Utrecht

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication (or other new use) have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors, and if not approved, may be further arbitrated by a Data Sharing Independent Review Panel. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the link below.
URL: https://www.amgen.com/datasharing

REFERENCES:
- [Derived] Cho SF, Lin L, Xing L, Li Y, Wen K, Yu T, Hsieh PA, Munshi N, Wahl J, Matthes K, Friedrich M, Arvedson T, Anderson KC, Tai YT. The immunomodulatory drugs lenalidomide and pomalidomide enhance the potency of AMG 701 in multiple myeloma preclinical models. Blood Adv. 2020 Sep 8;4(17):4195-4207. doi: 10.1182/bloodadvances.2020002524. PMID 32898244
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com